CLINICAL TRIAL: NCT04713566
Title: Comparative Clinical Effects of Salvadora Persica Oral Rinse And A Phenolic Commercial Mouth Wash On Human Oral Health
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Multan Medical And Dental College (Other)
Responsible Party: Principal Investigator, Dr. Aeeza Malik, Associate Professor, Multan Medical And Dental College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MMDC
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Plaque, Dental
Keywords: Dental plaque; Gingivitis; Miswak; Mouthwash
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): will be using Salvadora Persica oral rinse
  Interventions: Other: oral rinces
- Group B (Experimental): will be using Commercial Phenolic mouthwash.
  Interventions: Other: oral rinces

INTERVENTIONS:
Other: oral rinces — natural and commercial oral rinses were compared for efficacy

SUMMARY:
ABSTRACT:

OBJECTIVE: To compare the clinical effects of Salvadora persica (miswak) oral rinse and commercial Listerein mouth wash on oral health of socially deprived madrasa girls.

METHODS: Girls aged 18-22 years living permanently in a madrasa of Multan city will be recruited. Sample size and trial duration will be determined using the American Dental Association guidelines. Participants will be randomized into two interventional groups; A and B and will be either provided with Salvadora persica oral rinse and commercial Listerein mouth wash respectively. Pre, mid and post-intervention examinations will be executed by a blind and calibrated examiner using Turesky Quigley Hein Plaque and Loe and Silness Gingival indices. Statistical analysis will include descriptive statistics and two sample independent t-tests. The p-value of <0.05 will be considered significant at 95 % confidence level.

KEY WORDS: Dental plaque, Gingivitis, Miswak, Mouthwash

DETAILED DESCRIPTION:
Comparative clinical effects of Salvadora persica (miswak) oral rinse and commercial Listerein mouth wash will be studied on the oral health of socially deprived madrasa girls. Girls aged 18-22 years living permanently in a madrasa of Multan city will be recruited. Sample size and trial duration will be determined using the American Dental Association guidelines. Participants will be randomized into two interventional groups; A and B and were either provided with Salvadora persica oral rinse and commercial Listerein mouth wash respectively. Pre, mid and post-intervention examinations will be executed by a blind and calibrated examiner using Turesky Quigley Hein Plaque and Loe and Silness Gingival indices. Statistical analysis will include descriptive statistics and two sample independent t-tests. The p-value of <0.05 will be considered significant at 95 % confidence level.

ELIGIBILITY:
Exclusion Criteria:

* Participants/girls with any medical or dental disease,
* Participants/girls with any dental prosthesis,
* Those taken antibiotics in last 6 months,
* Those received any periodontal therapy in last 3 months

Inclusion Criteria:

*Participants with at least 10 sites of chronic mild gingivitis with bleeding on probing but not having periodontal pockets of greater than 3mm

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
plaque and gingivitis scores | 6 months
  Dental examination will be conducted at baseline, then after 3 and 6 months, that is, Pre-Interventional, Mid Intervention and Post-Interventional phases respectively. It will be executed on inclined chairs in day light using a sterilized dental mirror and CPITN (Community Periodontal Index of Treatment Need) probe. This probe has a ball ended tip with a diameter of 0.5mm. This probe have two coloured bands of 2mm graduations each, one at 3.5 to 5.5mm and second at 8.5 to 11.5mm. These bands determine the bleeding on probing which correspond to respective gingival score as per Loe and Silness Gingival index (1962)

CONTACTS AND LOCATIONS:
Overall Officials: Aeeza Malik, BDS, MDS, Principal Investigator — Multan Medical & Dental College
Locations (1):
- Aeeza Malik, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No